CLINICAL TRIAL: NCT06164704
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Efficacy and Safety of Verekitug (UPB-101) in Participants With Chronic Rhinosinusitis With Nasal Polyps on a Background of Nasal Corticosteroids (VIBRANT)
Brief Title: A Study to Investigate the Efficacy and Safety of Verekitug (UPB-101) in Participants With Chronic Rhinosinusitis With Nasal Polyps
Acronym: VIBRANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Upstream Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPB-CP-03; 2023-508231-31-00 (EU CTIS Number)
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: CRSwNP; Nasal Corticosteroids; VIBRANT; Nasal Polyps; Sinusitis; Paranasal Sinus Diseases; Nose Diseases; Respiratory Tract Diseases; Otorhinolaryngologic Diseases
MeSH Terms: conditions — Nasal Polyps; Sinusitis; Paranasal Sinus Diseases; Nose Diseases; Respiratory Tract Diseases; Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verekitug (UPB-101) (Experimental): Participants will be administered 0.5 milliliter (mL) of verekitug (UPB-101) formulated solution (containing 100 milligrams [mg] of verekitug [UPB-101]) subcutaneously, every 12 weeks for 24 weeks.
  Interventions: Drug: Verekitug (UPB-101)
- Matching placebo (Placebo Comparator): Participants will be administered verekitug (UPB-101) matching placebo solution, subcutaneously, every 12 weeks for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verekitug (UPB-101) — Verekitug (UPB-101) 0.5 mL of formulated solution (100 mg verekitug [UPB-101])
  Arms: Verekitug (UPB-101)
Drug: Placebo — Verekitug (UPB-101) matching placebo
  Arms: Matching placebo

SUMMARY:
The primary purpose of this study is to assess the effect of verekitug (UPB-101) on the endoscopically determined size and extend of nasal polyps in participants with chronic rhinosinusitis with nasal polyps (CRSwNP) and to assess the safety and tolerability of verekitug (UPB-101) compared to placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo controlled, parallel group study to assess the efficacy and safety of verekitug (UPB-101) administered subcutaneously (SC) in participants with CRSwNP on background therapy with stable dosage of intranasal corticosteroids (INCS). Approximately 70 participants will be randomized. Participants will receive verekitug (UPB-101) or placebo over a 24-week treatment period. In addition, this study consists of a 3 to 5-week Screening Period and a 4-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed, dated and received a copy of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form (ICF).
* Participant is aged 18 to 85 years of age (inclusive) at the time of signing the ICF.
* Participant has physician diagnosed CRSwNP for at least 6 months prior to Visit 1 that fulfills all of the following:

  * Severity consistent with need for surgery as defined by an endoscopic bilateral NPS of at least 5 out of 8 and a minimum score of 2 in each nasal cavity at Visit 1 based on central reading, as well as reconfirmed at Visit 2 based on local reading.
  * Average NCS greater than and equal to (>=) 2 over 14 days before Visit 2.
  * Ongoing symptoms of CRSwNP for at least 8 weeks prior to Visit 1 such as rhinorrhea and/or reduction in smell.
* Participant has at least one of the following:

  * In the 24 months prior to Visit 1, had a documented exacerbation of nasal polyposis requiring treatment with systemic corticosteroid.
  * A medical contraindication/intolerance to systemic corticosteroid.
  * Had prior surgery for NP (cannot be within 6 months prior to Visit 1
* Stable standard of care treatment for CRSwNP for at least 30 days prior to Visit 1.
* At Visit 2, at least 21 days of background mometasone furoate nasal spray (MFNS) (or equivalent) background therapy.
* >=70 percent (%) dosing compliance for MFNS (or equivalent) in the 14 days prior to Visit 2.
* Agrees to follow the required contraceptive techniques/methods
* Female or male participant agrees not to donate eggs or sperm, respectively, for a period of 120 days after the last dose of the study drug intervention or at the Final Visit, whichever occurs last

Exclusion Criteria:

* Has undergone any intranasal and/or sinus surgery (including polypectomy) within 6 months prior to Visit 1.
* Expected need, in the opinion of the Investigator, for NP surgery within 12 weeks of Visit 2.
* Comorbid asthma having forced expiratory volume in 1 second (FEV1) 50% or less of predicted normal at Visit 1.
* Conditions making participants non-evaluable at Visit 1 for the primary endpoint such as sino-nasal or sinus surgery changing the lateral wall structure of the nose, antrochoanal polyps, nasal septal deviation occluding at least one nostril, acute sinusitis, upper respiratory infection, ongoing rhinitis medicamentosa, fungal rhinosinusitis, nasal cavity benign or malignant tumors.
* Concurrent participation in a clinical study or has been treated with an investigational drug within 28 days or 5 half-lives, whichever is longer, prior to Visit 1.
* Previous exposure to verekitug (UPB-101) or known allergy/sensitivity to any of its excipients.
* Biologic therapy or systemic immunosuppressant to treat inflammatory disease or autoimmune disease within 6 months or 5 half-lives before Visit 1, whichever is longer, with the exception of oral c corticosteroids.
* Any vaccination within the Screening Period and treatment with a live (attenuated) vaccine within 12 weeks before Visit 2.
* Abnormal medical history, physical finding or safety finding and any clinical laboratory test result outside of the reference ranges that in the opinion of the Investigator may obscure the study data or interfere with the participant's safety. Participants with any clinically significant cardiac disease and/or ECG abnormality, in the opinion of the Investigator, obtained during the Screening Period should be excluded from the study.
* Allergic granulomatous angiitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis), Young's syndrome, Kartagener's syndrome or other dyskinetic ciliar syndromes, concomitant cystic fibrosis.
* Participant with comorbid asthma that also has a history or evidence of a clinically significant pulmonary condition (other than asthma).
* History of chronic alcohol or substance use disorder within 12 months prior to Visit 1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Nasal Polyp Score (NPS) at Week 24 | At Week 24
  Bilateral endoscopic NPS is a physician-reported scoring system to estimate the extent or severity of nasal polyps (NPs) based on assessments by nasal endoscopy. Each nostril is scored on a categorical scale of 0 to 4. The total score is the sum of the right and left scores (0-8). A higher score means severe disease.

SECONDARY OUTCOMES:
Change From Baseline in the Nasal Congestion Score (NCS) Evaluated by the Nasal Polyposis Symptom Diary (NPSD) at Week 24 | At Week 24
  Nasal congestion will be reported by participants daily, recalling nasal congestion severity over the previous 24 hours as none, mild, moderate, or severe (scores of 0, 1, 2, or 3, respectively). A higher score means worse outcome.
Change From Baseline in Opacification of Sinuses Measured by Lund Mackay Score (LMK) at Week 24 | At Week 24
  LMK score or sinus opacification score is a physician-reported quality staging system for evaluation of severity of NPs based on assessments of the sinuses by computer tomography (CT). CT scans will not be performed in Germany and Czechia. The LMK staging system assigns a value of 0, 1, or 2 to each of the following 5 sinuses: maxillary, anterior ethmoid, posterior ethmoid, frontal, and sphenoid where in 0=sinus is totally patent, 1=sinus is partially opacified, 2=sinus completely opacified; A higher score means severe disease.
Change From Baseline in Mean Difficulty With Sense of Smell (DSS) Evaluated by the NPSD at Week 24 | At Week 24
  Loss of smell based on participant-reported assessment of symptom severity of DSS, recalled over the past 24 hours. For the assessment, participants will be asked to assess their DSS for the previous day on a 4-point verbal scale of 0=none to 3=severe and record it in the electronic Diary. Higher daily DSS score indicates greater severity.
Percentage of Participants Requiring Systemic Corticosteroids or NP Surgery | Up to Week 24
  Percentage of participants requiring systemic corticosteroids or NP surgery will be recorded.
Time to First NP Surgery and/or Use of Systemic Corticosteroids for NP up to Week 24 | Up to Week 24
  Time to first NP surgery and/or use of systemic corticosteroids for NP will be recorded.
Change From Baseline in NPSD - Total Symptom Score (TSS) at Week 24 | At Week 24
  Participants will complete a NPSD each morning. Questions will be asked to report common symptoms of nasal polyposis and symptom impacts. Participants will report severity of each symptom and symptom impact at its worse using a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). Higher score indicates more severe symptoms.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | From Baseline up to Week 28
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Patel, MD, Study Director — Upstream Bio
Locations (41):
- United States (27):
  - Sensa Health LA (Sensa Health Clinical Research), Los Angeles, California
  - NewportNativeMD, Inc., Newport Beach, California
  - DaVinci, Research LLC, Roseville, California
  - Senta Clinic, San Diego, California
  - University of Missouri, Columbus, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Alfa Medical Research, Hollywood, Florida
  - Novaceut Clinical Research, Miami, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - IMIC Inc., Miami, Florida
  - University of South Florida, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - The University of Chicago, Chicago, Illinois
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Northwell Health/Division of Allergy and Immunology, Great Neck, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Spartanburg /Greer ENT & Allergy, Spartanburg, South Carolina
  - Orion Clinical Research, Austin, Texas
  - Alina Clinical Trials, LLC., Dallas, Texas
  - Ears Nose and Throat Associates of Texas, McKinney, Texas
  - Alamo Ent Associates, San Antonio, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington
  - Allergy, Asthma and Sinus Center, S.C., Greenfield, Wisconsin
- NZZ MUDr Pavel Navratil, Olomouc, Czech Republic, Czechia
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinik Muenster, Klinik fur Hals-, Nasen- und Ohrenheilkunde, Münster
  - Universitätsklinik Tuebingen, Tübingen
- Poland (5):
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Medyczne "All-Med" Badania Kliniczne spolka komandytowa, Krakow
  - Centrum Medyczne PROMED, Krakow
  - CENTRUM SŁUCHU I MOWY Sp. z o.o., Nadarzyn
  - Centrum Medyczne Lucyna Andrzej Dymek s.c, Strzelce Opolskie
- Spain (5):
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario de Jerez de la Frontera, Cadiz
  - Hospital Universitario Fundacion Jimenez Diaz (UAM-FJD) Consultas Externas Isaac Peral, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No